CLINICAL TRIAL: NCT05602155
Title: Comparison of Full-Weight and Partial-Weight-Bearing Patient Groups in Patients Over 65 Years of Age Who Underwent Proximal Femoral Nail Due to Intertrochanteric Fracture of the Femur
Brief Title: Partial Weight Bearing Proximal Femoral Nail Due to Intertrochanteric Fracture.
Acronym: randomized
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Duran Topak, Orthopaedic Clinical Assoc. Prof., Kahramanmaras Sutcu Imam University
Other Study IDs: 13.07.2018\16
Record Dates: First submitted 2022-10-18; First posted 2022-11-01 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Femur Intertrochanteric Fractures
Keywords: intertrochanteric fracture; elderly fractures; weight bearing
MeSH Terms: conditions — Hip Fractures | interventions — Partial Weight-Bearing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: weight bearing situation: patients with partial weight bearing after treatment
  Interventions: Procedure: Group 1; Procedure: Group 2
- Group 2: weight bearing: patients with full weight bearing after treatment
  Interventions: Procedure: Group 1; Procedure: Group 2

INTERVENTIONS:
Procedure: Group 1 — Even numbered patients will partial weight bearing after treatment,
  Other Names: partial weight bearing
Procedure: Group 2 — patients with odd numbers will walk with full weight bearing after treatment
  Other Names: full weight bearing

SUMMARY:
Femur intertrochanteric fractures (FITC) are one of the most common fractures of the lower extremity, caused by osteoporosis, caused by minor trauma in elderly patients. Today, it is successfully treated with proximal femoral nails (PFN) designed in different ways. After surgical fixation with PFN, patients are mobilized by placing full weight, but some complications can be seen due to the patients being osteoporotic. In this study, the investigators planned to investigate the effect of full weight bearing and partial weight bearing on complications, which were not previously described in the literature.

DETAILED DESCRIPTION:
Participants over the age of 60 who underwent PFN with the diagnosis of FITK were randomized (double-blinded consecutive full load on one patient and partial weight on one patient), and mobilized a group with full weight with the help of a walker after surgical fixation, and the other group with the help of a walker to give partial weight (balance). We planned to follow up his treatment prospectively. The compatibility of the groups will be evaluated by comparing the bone mineral density, calcium, alkaline phosphatase, phosphate, vitamin D levels and ages of the patients. Fracture types and post-treatment reduction quality of patients in both groups will be compared. We planned to compare the complication rates, Barthel Index and harris hip scores in the follow-up of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 65 years of age with intertrochanteric femoral fractures
2. Patients treated with proximal femoral nail
3. Patients able to walk before treatment
4. Patients who can be contacted

Exclusion Criteria:

1. Patients without regular follow-up for 1 year
2. Patients who do not walk before or after fracture
3. who have a neurological disease
4. Patients with partial hip replacement after fracture
5. Patients who cannot be contacted after treatment
6. Patients who died within 1 year after treatment

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — over 60 ages
Study Population: 1. Patients over 65 years of age who underwent proximal femoral nail due to femoral intertrochanteric fracture
Sampling Method: Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
demographic datas | August 2018
  Descriptive statistical data
comparison of groups | 1 year after surgery
  harris hip score: The Turkish version of the Harris hip score with adequate internal consistency (Cronbach's alpha, 0.70) and test-retest reliability (ICC = 0.91) was used for functional outcomes. It is evaluated with scores ranging from 0 to 100. The higher the score, the better the hip function.
comparison of groups | 6 month after operative treatment
  Barthel Index: The Turkish version of the Barthel index, which was developed by Mahoney and Barthel in 1965, and edited by Küçükdeveci et al., was used to evaluate the degree of independence of patients in activities of daily living. In this scale, where the possible score is between 0-100, the high score means that the patient is independent from other people and can run his own business; 0-20 points are defined as fully dependent, 21-61 points severely dependent, 62-90 points moderately dependent, 91-99 points mildly dependent, and 100 points fully independent
comparison of groups | At the beginning of the study
  age (year)
comparison of groups | before surgery
  Vit D (microgram\L)
comparison of groups | august 2022
  Complication (cut out, Z effect, infection, implant failure)
comparison of groups | On completion of the study, an average of 1 year
  Union time (week): Fracture union was defined radiologically as visible callus formation and reduction in pain in the groin.
comparison of groups | patient's last control date, at least 1 year later
  Following time (month): The time elapsed between the date the patient came for the last control and the first application

CONTACTS AND LOCATIONS:
Overall Officials: Ökkeş Bilal, 3., Study Chair — Assistant researcher
Locations (1):
- Duran Topak, Kahramanmaraş, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Patients over the age of 60 who underwent PFN with the diagnosis of FITK were randomized (double-blinded consecutive full load on one patient and partial weight on one patient), and mobilized a group with full weight with the help of a walker after surgical fixation, and the other group with the help of a walker to give partial weight (balance). We planned to follow up his treatment prospectively. The compatibility of the groups will be evaluated by comparing the bone mineral density, calcium, alkaline phosphatase, phosphate, vitamin D levels and ages of the patients. Fracture types and post-treatment reduction quality of patients in both groups will be compared. We planned to compare the complication rates and harris hip scores in the follow-up of the patients.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5 years
Access Criteria: for researchers

REFERENCES:
- [Result] Kucukdeveci AA, Yavuzer G, Tennant A, Suldur N, Sonel B, Arasil T. Adaptation of the modified Barthel Index for use in physical medicine and rehabilitation in Turkey. Scand J Rehabil Med. 2000 Jun;32(2):87-92. PMID 10853723
- [Result] Jensen JS. Classification of trochanteric fractures. Acta Orthop Scand. 1980 Oct;51(5):803-10. doi: 10.3109/17453678008990877. PMID 7468173
- See also: Barthel index — https://pubmed.ncbi.nlm.nih.gov/10853723/
- See also: Fracture classification — https://pubmed.ncbi.nlm.nih.gov/7468173/